CLINICAL TRIAL: NCT01205165
Title: An Open Label, Multicenter Phase IV Study of Adefovir Dipivoxil in Korean Patients With Chronic Hepatitis B (CHB)
Brief Title: An Open Label, Multi Centre Phase IV Study of Adefovir Dipivoxil in Korean Patients With Chronic Hepatitis B (CHB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103814
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adefovir Dipivoxil 10mg (Experimental): All enrolled subject were enrolled to adefovir dipivoxil 10mg arm.
  Interventions: Drug: Adefor dipivoxil

INTERVENTIONS:
Drug: Adefor dipivoxil — All enrolled subjects were enrolled to adefovir dipivoxil arm.

SUMMARY:
Objective(s) The primary study objective is to assess the antiviral effect of 12 weeks of adefovir dipivoxil treatment in Korean patients with chronic hepatitis B and compensated liver disease. The secondary study objectives are to assess the antiviral effect, clinical benefit and safety of 52 weeks of adefovir dipivoxil treatment.

Endpoint(s) The primary efficacy endpoint is "Mean log10 reduction in serum HBV DNA level from baseline to Week 12".

The secondary efficacy endpoints include (a) the proportion of patients achieving serum ALT normalization at Week 52, (b) other assessments of antiviral effects (the proportion of patients achieving HBV DNA no less than 300 copies per mL at Week 52), (c)HBeAg loss, HBeAg seroconversion, HBsAg loss and HBsAg seroconversion, (d)the proportion of patients achieving serum ALT normalization at Week 12.

Study Design This is an open label, multi centre phase IV study for Korean patients with chronic hepatitis B and compensated liver disease, assessing the antiviral effect of 12 weeks treatment of Adefovir dipivoxil as a primary objective and antiviral effect, clinical benefit and safety of 52 weeks treatment as secondary objectives.

Patients will be screened for eligibility criteria and the baseline visit for the treatment initiation should occur no more than 4 weeks after screening. Total treatment period will be 52 weeks and patients will return to the clinic for assessments as scheduled during treatment period. After the 52 week study period, it is likely that the patient will benefit from continued treatment with commercial adefovir. If in the investigator's clinical judgement this is the case, the investigator should ensure that a routine prescription is available in a timely manner, and that no unnecessary interruption in treatment occurs.

Study Population A minimum of 100 male or female Korean patients more than 18 years of age with HBeAg positive chronic hepatitis B and compensated liver disease who meet the eligibility criteria will be enrolled.

Study Assessments and Procedures

Potential patients will be screened prior to study entry and eligible patients who have given their consent will have further baseline assessments. Following the screening, the first doses of study medications will be given at baseline and patients will return to the clinic for assessment as scheduled during treatment period. Patients who discontinue treatment prematurely will be followed up every 4 weeks for 12 weeks following the withdrawal visit. The following key assessment and or measurement will be made at one or more visits during the study. (See section 14.1 Appendix 1. Time and event schedule):

* Pregnancy test (females of child-bearing potential only)
* Haematology and serum chemistry profile including prothrombin time(PT) and AFP
* HBV DNA (Roche COBAS AMPLICOR HBV MONITOR Test, LLOD 300 copies per ml)
* Hepatitis B markers: HBeAg(Anti HBe will be tested if HBeAg is negative), HBsAg(Anti HBs will be tested if HBsAg is negative) Investigational Product(s) Adefovir dipivoxil 10mg tablets will be supplied by GlaxoSmithKline and presented as a white to off white, round tablets, packaged in the bottle containing 30 tablets

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Age more than 18 years
2. HBV Serology Presence of HBsAg for at least 6 months Presence of HBeAg at the time of screening Positive HBV DNA plasma assay with screening value at the time of screening

4. Evidence of at least one elevated serum alanine amonotransferase (ALT) levels greater than 2 times (inclusive) the upper limit of the normal range (ULN) in the previous 6 months.

serum ALT levels greater than 2 times (inclusive) the ULN at screening visit. 5. Availability and willingness of subject to provide written informed consent.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Use of immunosuppressive therapy requiring use of more than 5mg of prednisone(or equivalent) per day, immunomodulatory therapy (including interferon or thymosin ) or systemic cytotoxic agents within previous 6 months or during the study
2. Previous or current lamivudine or adefovir dipivoxil therapy or antiviral therapy with agents demonstrating potential anti-HBV activity
3. Clinical signs of decompensated liver disease at screening according to the protocol
4. Serum creatinine over 1.5mg per dL
5. Alanine aminotransferase (ALT) over 10 times ULN at screening or history of acute exacerbation leading to transient decompensation
6. Serum Amylase and/or lipase over 2 times ULN
7. Inadequate haematological function
8. Anti-HBe or Anti-HBs positive subjects
9. Hepatocellular carcinoma as evidenced by the protocol
10. Documented evidence of active liver disease
11. Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include any uncontrolled clinically significant renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders or cancer.
12. Active alcohol or drug abuse or history of alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
13. Planned for liver transplantation or previous liver transplantation
14. Receipt of any investigational drug within within 3 months prior to screening.
15. Therapy with nephrotoxic drugs or competitors of renal excretion within 2 months prior to study screening or the expectation that patient will receive any of these during the course of the study.
16. History of hypersensitivity to nucleoside and/or nucleotide analogues.
17. Inability to comply with study requirements as determined by the study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-12-17 (Actual); Primary Completion 2006-04-28 (Actual); Study Completion 2006-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in participants with chronic hepatitis B and compensated liver disease, at 5 sites in Korea. It was conducted from 01 December 2004 to 28 April 2006.
Pre-assignment Details: Of the total 140 participants which were screened only 104 participants were randomized to the study.
Groups:
- Adefovir Dipivoxil 10mg: The eligible participants received open label treatment of 10 milligram (mg) Adefovir dipivoxil, orally once daily for 52-weeks
Period: Overall Study
Arm/Group | Adefovir Dipivoxil 10mg
Started | 104
Completed | 102
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Adefovir Dipivoxil 10mg: The eligible participants received open label treatment of 10 mg Adefovir dipivoxil, orally once daily for 52-weeks
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 83
Region of Enrollment [Number; unit: Participants]
  Korea | 104

OUTCOME MEASURES:

1. Primary Outcome: Mean Log 10 Reduction in Serum Hepatitis B Virus (HBV), Deoxyribonucleic Acid (DNA) Level From Baseline to Week 12
Description: HBV DNA was tested with Roche Cobas Amplicor HBV monitor test, where the lower limit of detection was 300 copies/milliliter (mL), at baseline and other study visits. The mean log 10 reduction in serum HBV DNA level from baseline to week 12 was calculated as the week 12 value minus the baseline value. Baseline was the Day 1 for the study, when participant received study drug. Log 10 reduction implied reduced viral load.
Time Frame: Baseline (Day 1) and Week 12
Population: Intent to treat (ITT). All participants regardless of whether or not the participant completed the planned duration of the study were analyzed with no data exclusions.
Measure: Mean (Standard Deviation); unit: Log10 (copies/mL)
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Log10 (copies/mL) | -3.39 (1.50)
Statistical Analysis 1: Comparison: Adefovir Dipivoxil 10mg; Baseline and Week 12; Test type: Superiority or Other; p = 0.00000, Wilcoxon signed rank test — P-value is calculated from Wilcoxon signed rank test to compare difference between baseline and week12

2. Secondary Outcome: Number of Participants Achieving Alanine Aminotransferase (ALT) Normalization at Week 52
Description: ALT normalization was defined as measurement less than or equal to the upper limit of the normal range. Only those set of participants with a baseline ALT value above the upper limit of the normal range was included in this analysis. The normal range for ALT is 7 to 43 Units/Liter.
Time Frame: At week 52
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants | 83

3. Secondary Outcome: Number of Participants Achieving Virological Response at Week 52
Description: Virological response was defined as HBV DNA level < 300 copies/ml in serum. The number of participants achieving these DNA levels were reported.
Time Frame: At Week 52
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants | 34

4. Secondary Outcome: HBV DNA Levels at Each Collection Timepoint Through Week 52
Description: Serum HBV DNA at different timepoints namely Baseline, Week 4, week 8, week 12, week 20, week 28, week 36, week 44 and week 52 were reported. The HBV DNA copies in the serum were reported in multiples of log 10 copies per mL, detected using Roche COBAS AMPLICOR HBV monitor.
Time Frame: Week 4, week 8, week 12, week 20, week 28, week 36, week 44 and week 52
Population: ITT population. Only those participants available at the specified timepoints were analyzed
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
log 10 copies/mL
  Week 4 | 5.59 (0.83)
  Week 8 | 4.96 (0.99)
  Week 12 | 4.56 (1.13)
  Week 20 | 3.97 (1.13)
  Week 28: number analyzed (Participants) | 103
  Week 28 | 3.92 (1.14)
  Week 36: number analyzed (Participants) | 103
  Week 36 | 3.78 (1.15)
  Week 44: number analyzed (Participants) | 102
  Week 44 | 3.63 (1.13)
  Week 52: number analyzed (Participants) | 101
  Week 52 | 3.66 (1.18)

5. Secondary Outcome: Number of Participants With Hepatitis B e Viral Protein (HBeAg) Loss, HBeAg Seroconversion, Hepatitis B Virus Surface Antigen (HBsAg) Loss and HBsAg Seroconversion at Week 52
Description: The HBeAg loss, defined as the number of participants with an undetectable level of serum HBeAg. The percentage of participants with a HBeAg seroconversion, defined as an undetectable level of serum HBeAg and a detectable level of serum hepatitis B e antibody (HBeAb) at Week 52. The number of participants with HBsAg loss was defined as an undetectable level of serum HBsAg; and those participants with HBsAg seroconversion were defined as an undetectable level of serum HBsAg and a detectable level of serum HBsAb. All these participant were reported at week 52. Only the subset of participants, with above parameters detectable at baseline were included and for participants with post-baseline values missing were considered as non-responders.
Time Frame: Week 52
Population: ITT population. Only the subset of participants with HBeAg and HBsAg positive at baseline (Day 1) was included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants
  HbeAg loss: number analyzed (Participants) | 103
  HbeAg loss | 19
  HbeAg seroconversion: number analyzed (Participants) | 103
  HbeAg seroconversion | 10
  HbsAg loss | 0
  HbsAg seroconversion | 0

6. Secondary Outcome: Number of Participants Achieving ALT Normalization at Week 12
Description: ALT normalization was defined as measurement less than or equal to the upper limit of the normal range. The normal range for ALT is 7-43 Units/Liter. Only those set of participants with a baseline ALT value above the upper limit of the normal range were included in this analysis, done at week 12.
Time Frame: at Week 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants | 50

7. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAEs)
Description: AE is defined as, any untoward medical occurrence in a participant or clinical investigation, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that at any dose, results in death; is life threatening; requires hospitalization or prolongation of hospitalization; results in disability or incapacity, is a congenital anomaly/birth defect or requires medical intervention.
Time Frame: From treatment initiation (Week 0) to follow-up (up to 52 weeks)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants
  All SAE's | 2
  All AE's | 43
  AEs related to study drug | 6

8. Secondary Outcome: Number of Participants With Shift From Baseline Hematology Parameters at Week 12 and Week 52
Description: The data for hematology parameters was summarized for Hemoglobin, Red blood cells (RBC), Platelets, Neutrophils, Lymphocytes, Monocytes, and Eosinophil as per the scheduled assessments and also according to maximum grade common terminology criteria (CTC) toxicity grade. The data for number of participants with shift in grade for hematology parameters at Week 12 and Week 52 were reported.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants
  Hemoglobin, Low to Normal, Week 12 | 0
  Hemoglobin, Low to High, Week 12 | 0
  Hemoglobin, High to Low, Week 12 | 0
  Hemoglobin, High to Normal, Week 12 | 3
  Hemoglobin, Normal to Low, Week 12 | 1
  Hemoglobin, Normal to High Week 12 | 3
  Hemoglobin, Low to Normal, Week 52 | 3
  Hemoglobin, Low to High, Week 52 | 0
  Hemoglobin, High to Low, Week 52 | 0
  Hemoglobin, High to Normal, Week 52 | 0
  Hemoglobin, Normal to Low, Week 52 | 1
  Hemoglobin, Normal to High Week 52 | 4
  RBC, Low to Normal, Week 12 | 4
  RBC, Low to High, Week 12 | 0
  RBC, High to Low, Week 12 | 0
  RBC, High to Normal, Week 12 | 0
  RBC, Normal to Low, Week 12 | 1
  RBC, Normal to High Week 12 | 2
  RBC, Low to Normal, Week 52 | 3
  RBC, Low to High, Week 52 | 0
  RBC, High to Low, Week 52 | 0
  RBC, High to Normal, Week 52 | 0
  RBC, Normal to Low, Week 52 | 1
  RBC, Normal to High Week 52 | 4
  Platelets, Low to Normal, Week 12 | 5
  Platelets, Low to High, Week 12 | 0
  Platelets, High to Low, Week 12 | 0
  Platelets, High to Normal, Week 12 | 0
  Platelets, Normal to Low, Week 12 | 2
  Platelet, Normal to High, Week 12 | 0
  Platelets, Low to Normal, Week 52 | 5
  Platelets, Low to High, Week 52 | 0
  Platelets, High to Low, Week 52 | 0
  Platelets, High to Normal, Week 52 | 0
  Platelet, Normal to Low, Week 52 | 0
  Platelets, Normal to High, Week 52 | 0
  Total WBC, Low to Normal, Week 12 | 10
  Total WBC, Low to High, Week 12 | 0
  Total WBC, High to Low, Week 12 | 0
  Total WBC, High to Normal, Week 12 | 0
  Total WBC, Normal to Low, Week 12 | 1
  Total WBC, Normal to High Week 12 | 1
  Total WBC, Low to Normal, Week 52 | 12
  Total WBC, Low to High, Week 52 | 0
  Total WBC, High to Low, Week 52 | 0
  Total WBC, High to Normal, Week 52 | 0
  Total WBC, Normal to Low, Week 52 | 3
  Total WBC, Normal to High, Week 52 | 3
  Neutrophils, Low to Normal, Week 12 | 11
  Neutrophils, Low to High, Week 12 | 0
  Neutrophils, High to Low, Week 12 | 0
  Neutrophils, High to Normal, Week 12 | 1
  Neutrophils, Normal to Low, Week 12 | 6
  Neutrophils, Normal to High, Week 12 | 0
  Neutrophils, Low to Normal, Week 52 | 14
  Neutrophils, Low to High, Week 52 | 0
  Neutrophils, High to Low, Week 52 | 0
  Neutrophils, High to Normal, Week 52 | 1
  Neutrophils, Normal to Low, Week 52 | 3
  Neutrophils, Normal to High, Week 52 | 2
  Lymphocytes, Low to Normal, Week 12 | 1
  Lymphocytes, Low to High, Week 12 | 0
  Lymphocytes, High to Low, Week 12 | 0
  Lymphocytes, High to Normal, Week 12 | 9
  Lymphocytes, Normal to Low, Week 12 | 1
  Lymphocytes, Normal to High Week 12 | 6
  Lymphocytes, Low to Normal, Week 52 | 1
  Lymphocytes, Low to High, Week 52 | 0
  Lymphocytes, High to Low, Week 52 | 0
  Lymphocytes, High to Normal, Week 52 | 12
  Lymphocytes, Normal to Low, Week 52 | 4
  Lymphocytes, Normal to High, Week 52 | 1
  Monocytes, Low to Normal, Week 12 | 0
  Monocytes, Low to High, Week 12 | 0
  Monocytes, High to Low, Week 12 | 0
  Monocytes, High to Normal, Week 12 | 15
  Monocytes, Normal to Low, Week 12 | 0
  Monocytes, Normal to High, Week 12 | 1
  Monocytes, Low to Normal, Week 52 | 0
  Monocytes, Low to High, Week 52 | 0
  Monocytes, High to Low, Week 52 | 0
  Monocytes, High to Normal, Week 52 | 16
  Monocytes, Normal to Low, Week 52 | 0
  Monocytes, Normal to High, Week 52 | 1
  Eosinophils, Low to Normal, Week 12 | 2
  Eosinophils, Low to High, Week 12 | 0
  Eosinophils, High to Low, Week 12 | 0
  Eosinophils, High to Normal, Week 12 | 3
  Eosinophils, Normal to Low, Week 12 | 1
  Eosinophils, Normal to High Week 12 | 1
  Eosinophils, Low to Normal, Week 52 | 2
  Eosinophils, Low to High, Week 52 | 0
  Eosinophils, High to Normal, Week 52 | 5
  Eosinophils, High to Low, Week 52 | 0
  Eosinophils, Normal to High, Week 52 | 4
  Eosinophils, Normal to Low, Week 52 | 2

9. Secondary Outcome: Number of Participants With Shift From Baseline Clinical Chemistry Parameters at Week 12 and Week 52
Description: The data for clinical chemical parameters namely sodium, potassium, calcium, phosphorus, total protein, albumin, amylase, creatinine phospho kinase, creatinine, blood urea nitrogen, total bilirubin, alkaline phosphatase, aspartate transaminase, alanine transaminase, and prothrombin time as per the scheduled assessments and also according to maximum CTC toxicity grade was reported. The data for number of participants with shift in grade for clinical chemistry parameters at Week 12 and Week 52 were reported.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: ITT population. Only those participants available at the specified time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Participants
  Sodium, Low to Normal, Week 12 | 0
  Sodium, Low to High, Week 12 | 0
  Sodium, High to Low, Week 12 | 0
  Sodium, Normal to Low, Week 12 | 2
  Sodium, High to Normal, Week 12 | 0
  Sodium, Normal to High, Week 12 | 1
  Sodium, Low to Normal, Week 52 | 0
  Sodium, Low to High, Week 52 | 0
  Sodium, High to Low, Week 52 | 0
  Sodium, High to Normal, Week 52 | 0
  Sodium, Normal to Low, Week 52 | 0
  Sodium, Normal to High, Week 52 | 2
  Potassium, Low to Normal, Week 12 | 1
  Potassium, Low to High, Week 12 | 0
  Potassium, High to Low, Week 12 | 0
  Potassium, High to Normal, Week 12 | 0
  Potassium, Normal to Low, Week 12 | 0
  Potassium, Normal to High, Week 12 | 1
  Potassium, Low to Normal, Week 52 | 1
  Potassium, Low to High, Week 52 | 0
  Potassium, High to Low, Week 52 | 0
  Potassium, High to Normal, Week 52 | 0
  Potassium, Normal to Low, Week 52 | 1
  Potassium, Normal to High, Week 52 | 0
  Calcium, Low to Normal, Week 12 | 1
  Calcium, Low to High, Week 12 | 0
  Calcium, High to Low, Week 12 | 0
  Calcium, High to Normal, Week 12 | 3
  Calcium, Normal to Low, Week 12 | 1
  Calcium, Normal to High, Week 12 | 2
  Calcium, Low to Normal, Week 52 | 1
  Calcium, Low to High, Week 52 | 0
  Calcium, High to Low, Week 52 | 0
  Calcium, High to Normal, Week 52 | 2
  Calcium, Normal to Low, Week 52 | 2
  Calcium, Normal to High, Week 52 | 0
  Phosphorus, Low to Normal, Week 12 | 4
  Phosphorus, Low to High, Week 12 | 0
  Phosphorus, High to Low, Week 12 | 0
  Phosphorus, High to Normal, Week 12 | 3
  Phosphorus, Normal to Low, Week 12 | 0
  Phosphorus, Normal to High, Week 12 | 3
  Phosphorus, Low to Normal, Week 52 | 4
  Phosphorus, Low to High, Week 52 | 0
  Phosphorus, High to Low, Week 52 | 0
  Phosphorus, High to Normal, Week 52 | 1
  Phosphorus, Normal to Low, Week 52 | 1
  Phosphorus, Normal to High, Week 52 | 1
  Total Protein, Low to Normal, Week 12 | 0
  Total Protein, Low to High, Week 12 | 0
  Total Protein, High to Low, Week 12 | 0
  Total Protein, High to Normal, Week 12 | 1
  Total Protein, Normal to Low, Week 12 | 0
  Total Protein, Normal to High, Week 12 | 3
  Total Protein, Low to Normal, Week 52 | 0
  Total Protein, Low to High, Week 52 | 0
  Total Protein, High to Low, Week 52 | 0
  Total Protein, High to Normal, Week 52 | 0
  Total Protein, Normal to Low, Week 52 | 0
  Total Protein, Normal to High, Week 52 | 4
  Amylase, Low to Normal, Week 12 | 0
  Amylase, Low to High, Week 12 | 0
  Amylase, High to Low, Week 12 | 0
  Amylase, High to Normal, Week 12 | 6
  Amylase, Normal to Low, Week 12 | 0
  Amylase, Normal to High, Week 12 | 3
  Amylase, Low to Normal, Week 52 | 0
  Amylase, Low to High, Week 52 | 0
  Amylase, High to Low, Week 52 | 0
  Amylase, High to Normal, Week 52 | 6
  Amylase, Normal to Low, Week 52 | 0
  Amylase, Normal to High, Week 52 | 2
  Creatinine phosphokinase, Low to Normal, Week 12 | 1
  Creatinine phosphokinase, Low to High, Week 12 | 0
  Creatinine phosphokinase, High to Low, Week 12 | 0
  Creatinine phosphokinase, High to Normal, Week 12 | 5
  Creatinine phosphokinase, Normal to Low, Week 12 | 0
  Creatinine phosphokinase, Normal to High, Week 12 | 2
  Creatinine phosphokinase, Low to Normal, Week 52 | 1
  Creatinine phosphokinase, Low to High, Week 52 | 0
  Creatinine phosphokinase, High to Low, Week 52 | 0
  Creatinine phosphokinase, High to Normal, Week 52 | 5
  Creatinine phosphokinase, Normal to Low, Week 52 | 0
  Creatinine phosphokinase, Normal to High, Week 52 | 3
  Creatinine, Low to Normal, Week 12 | 0
  Creatinine, Low to High, Week 12 | 0
  Creatinine, High to Low, Week 12 | 0
  Creatinine, High to Normal, Week 12 | 0
  Creatinine, Normal to Low, Week 12 | 0
  Creatinine, Normal to High, Week 12 | 2
  Creatinine, Low to Normal, Week 52 | 0
  Creatinine, Low to High, Week 52 | 0
  Creatinine, High to Low, Week 52 | 0
  Creatinine, High to Normal, Week 52 | 0
  Creatinine, Normal to Low, Week 52 | 0
  Creatinine, Normal to High, Week 52 | 3
  Blood urea nitrogen, Low to Normal, Week 12 | 7
  Blood urea nitrogen, Low to High, Week 12 | 0
  Blood urea nitrogen, High to Low, Week 12 | 0
  Blood urea nitrogen, High to Normal, Week 12 | 1
  Blood urea nitrogen, Normal to Low, Week 12 | 1
  Blood urea nitrogen, Normal to High, Week 12 | 0
  Blood urea nitrogen, Low to Normal, Week 52 | 10
  Blood urea nitrogen, Low to High, Week 52 | 0
  Blood urea nitrogen, High to Low, Week 52 | 0
  Blood urea nitrogen, High to Normal, Week 52 | 1
  Blood urea nitrogen, Normal to Low, Week 52 | 3
  Blood urea nitrogen, Normal to High, Week 52 | 0
  Total bilirubin, Low to Normal, Week 12 | 0
  Total bilirubin, Low to High, Week 12 | 0
  Total bilirubin, High to Low, Week 12 | 0
  Total bilirubin, High to Normal, Week 12 | 7
  Total bilirubin, Normal to Low, Week 12 | 0
  Total bilirubin, Low to Normal, Week 52 | 0
  Total bilirubin, Low to High, Week 52 | 0
  Total bilirubin, High to Low, Week 52 | 0
  Total bilirubin, High to Normal, Week 52 | 5
  Total bilirubin, Normal to Low, Week 52 | 0
  Total bilirubin, Normal to High, Week 52 | 9
  Alkaline phosphatase, Low to Normal, Week 12 | 0
  Alkaline phosphatase, Low to High, Week 12 | 0
  Alkaline phosphatase, High to Low, Week 12 | 0
  Alkaline phosphatase, High to Normal, Week 12 | 5
  Alkaline phosphatase, Normal to Low, Week 12 | 3
  Alkaline phosphatase, Normal to High, Week 12 | 2
  Alkaline phosphatase, Low to Normal, Week 52 | 0
  Alkaline phosphatase, Low to High, Week 52 | 0
  Alkaline phosphatase, High to Low, Week 52 | 0
  Alkaline phosphatase, High to Normal, Week 52 | 8
  Alkaline phosphatase, Normal to Low, Week 52 | 2
  Alkaline phosphatase, Normal to High, Week 52 | 1
  Prothrombin Time, Low to Normal, Week 12 | 1
  Prothrombin Time, Low to High, Week 12 | 0
  Prothrombin Time, High to Low, Week 12 | 0
  Prothrombin Time, High to Normal, Week 12 | 5
  Prothrombin Time, Normal to Low, Week 12 | 1
  Prothrombin Time, Normal to High, Week 12 | 6
  Prothrombin Time, Low to Normal, Week 52 | 2
  Prothrombin Time, Low to High, Week 52 | 0
  Prothrombin Time, High to Low, Week 52 | 0
  Prothrombin Time, High to Normal, Week 52 | 6
  Prothrombin Time, Normal to Low, Week 52 | 6
  Prothrombin Time, Normal to High, Week 52 | 2

10. Secondary Outcome: Mean Log 10 Reduction in Serum HBV DNA Level From Baseline to Week 52
Description: HBV DNA was tested with Roche Cobas Amplicor HBV monitor test, HBV DNA was tested with Roche Cobas Amplicor HBV monitor test, Lower Limit of Detection 300 copies/mL), at baseline and other study visits. The mean log 10 reduction in serum HBV DNA level from baseline to Week 52 was calculated as the Week 52 value minus the baseline value. Baseline was the Day 1 for the study when participant received study drug. Log 10 reduction implied reduced viral load
Time Frame: Baseline (Day 1) and Week 52
Population: ITT population
Measure: Mean (Standard Deviation); unit: Log10 (copies/mL)
Arm/Group | Adefovir Dipivoxil 10mg
Number analyzed (Participants) | 104
Log10 (copies/mL) | -4.32 (1.56)

ADVERSE EVENTS:
Time Frame: From treatment initiation (Week 0) to follow-up (up to 52 weeks)
Description: ITT population
Arm/Group | Adefovir Dipivoxil 10mg
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 2/104
Other Adverse Events (participants affected / at risk) | 16/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil 10mg (N=104)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Ascites (Hepatobiliary disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil 10mg (N=104)
Fatigue (General disorders) | 9
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.